CLINICAL TRIAL: NCT02746159
Title: A Prospective, Multicenter, Single Arm Real-World Registry Investigating the Clinical Use and Safety of the Lutonix Drug Coated Balloon PTA Catheter for Treatment of Dysfunctional Native and Synthetic AV Fistulae
Brief Title: Lutonix® Global AV Registry Investigating Lutonix Drug Coated Balloon for Treatment of Native and Synthetic AV Fistulae
Acronym: AVR
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: CL0026-01
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2019-08

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Lutonix 035 Drug Coated Balloon PTA Catheter, Model 9004

SUMMARY:
The purpose of this Registry is to enroll patients presenting with clinical and hemodynamic abnormalities in native or synthetic (grafts) arteriovenous (AV) fistulae located in the arm. Subjects will be treated with the Lutonix DCB carrying the CE Mark per current IFU and followed clinically for a minimum of 12 months.

DETAILED DESCRIPTION:
This post market registry is intended to demonstrate safety and assess the clinical use and outcomes of the Lutonix DCB in a heterogeneous patient population with dysfunctional native or synthetic AV fistulae in real world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-breastfeeding female ≥18 years of age;
2. Patient is willing to provide informed consent, and is willing to comply with the protocol-required follow up visits;
3. Native or synthetic (grafts) arteriovenous fistula located in the arm, including central veins, presenting with any clinical, physiological or hemodynamic abnormalities warranting angiographic imaging as defined in the K/DOQI guidelines; and
4. Lesion(s) can be treated with available Lutonix DCB device size matrix per current IFU.

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

1. Patient is currently participating in an investigational drug or device study which has not yet reached its primary endpoint or was previously enrolled into this registry (i.e. Lutonix Global AV registry).
2. Patient has a non-controllable allergy to contrast; or
3. Patient has another medical condition that, which in the opinion of the Investigator, may confound the data interpretation of is associated with a life expectancy insufficient to allow for completion of patient registry procedure and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients presenting with clinical and hemodynamic abnormalities in native or synthetic (grafts) arteriovenous (AV) fistulae located in the arm.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2019-03-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with freedom from any serious adverse event(s) involving the AV access circuit | 30 days.
  Primary safety events include any serious adverse event(s) involving the AV access circuit
Proportion of subjects with target lesion primary patency | 6 Months
  Defined as the interval following index procedure until clinically-driven reintervention of the target lesion or access thrombosis, through 6 months.
  Clinically-driven reintervention is defined as a lesion that has ≥50% stenosis and at least one clinical, physiological or hemodynamic abnormality attributable to the stenosis defined in the K/DOQI guidelines.

SECONDARY OUTCOMES:
Proportion of subjects with access circuit primary patency at 3, 6, and 12 months | 12 months
  Interval following intervention until the next access circuit thrombosis or repeated intervention. Ends with treatment of a lesion anywhere within the access circuit.
Proportion of Subjects withTarget Lesion Primary Patency (TLPP) | 12 months
  Target Lesion Primary Patency (TLPP) is defined as the interval following index procedure intervention until clinically driven reintervention of the target lesion or access thrombosis.
Proportion of Subjects with Abandonment of permanent access in the index extremity | 12 months
  The arteriovenous fistula / access circuit is considered abandoned when it is no longer being used for dialysis because the access was not functioning.
Proportion of Subjects with Device Success | 12 Months
  Successful delivery to the target lesion, deployment, and retrieval at index procedure. If a device is inserted into the subject but not used due to user error (e.g. inappropriate balloon length or transit time too long), this device will not be included in the device success assessment.
Proportion of Subjects with Procedural Success | 12 Months
  At least one indicator of hemodynamic success (e.g., physical examination with restoration of a thrill, direct measurement of flow) in the absence of peri-procedural (index procedure and through hospital stay) Serious Adverse Device Effects (SADEs).
Proportion of Subjects with Clinical Success | 12 Months
  The resumption of dialysis for at least one session after the index procedure.
Rate of device and procedure related adverse events | 12 months
  Freedom from device-related or procedure-related serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karnabatidis, MD, PhD, Principal Investigator — University Hospital of Patras, Radiology Department
Locations (26):
- LKH Graz, Graz, Austria
- France (3):
  - Clinique du Pré, Le Mans
  - Clinique Les Fontaines, Melun
  - Institut Montsouris, Paris
- Germany (2):
  - Uniklinik Giessen und Marburg, Giessen
  - Universitätsklinikum Jena, Jena
- University Hospital of Patras, Pátrai, Greece
- Italy (4):
  - Azienda Ospedaliera Di Pisa - Ospedale Cisanello, Pisa
  - Casa Di Cura Maria Rosaria, Pompei
  - San Giovanni Bosco, Torino
  - University of Insubria, Varese
- Klinika Chirurgii Naczyniowej University Hospital nr 1, Lublin, Poland
- Portugal (2):
  - Hospital da Cruz Vermelha, Lisbon
  - NephroCare Portugal, S.A. NephroCare Lumia, Lisbon
- King Abdullah International Medical Research Center, Riyadh, Saudi Arabia
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Ospedale Regionale di Lugano, Lugano, Switzerland
- Taiwan (4):
  - Buddhist Dalin Tzuchi hospital, Dalin
  - Chang-Gung Memorial Hospital, Linkou District
  - Hsin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Tzu Chi Hospital, Taipei
- Ankara Baskent University, Ankara, Turkey (Türkiye)
- United Kingdom (3):
  - Lister Hospital, Leicester
  - Barts and The Royal London Hospital, London
  - Royal Berkshire hospital, Reading

IPD SHARING:
Plan to Share IPD: No